CLINICAL TRIAL: NCT04824742
Title: A Prospective Randomized Controlled Study of Neoadjuvant PDT in the Treatment of Cholangiocarcinoma
Brief Title: Neoadjuvant PDT in the Treatment of Cholangiocarcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020ZDLSF04-08
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cholangiocarcinoma Resectable
Keywords: Cholangiocarcinoma,Neoadjuvant therapy,Photodynamic therapy
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant PDT + radical surgery (Experimental): Photodynamic therapy for neoadjuvant treatment of cholangiocarcinoma
  Interventions: Procedure: Neoadjuvant PDT + radical surgery
- radical surgery (Active Comparator): Patients with cholangiocarcinoma undergo radical surgical resection
  Interventions: Procedure: Radical surgery

INTERVENTIONS:
Procedure: Neoadjuvant PDT + radical surgery — Patients with cholangiocarcinoma will undergo radical surgery after photodynamic therapy
  Arms: neoadjuvant PDT + radical surgery
Procedure: Radical surgery — Patients with cholangiocarcinoma will only receive radical surgery
  Arms: radical surgery

SUMMARY:
For patients with locally advanced cholangiocarcinoma with resectable margins, patients who meet the selection criteria are randomly divided into two groups A and B. Group A: neoadjuvant PDT therapy combined with radical surgery; Group B: radical surgery. This study aims to explore the clinical effectiveness and safety of neoadjuvant photodynamic therapy for cholangiocarcinoma, as well as its role in destroying local tumors and enhancing systemic inflammation.

DETAILED DESCRIPTION:
The average 5-year survival rate of patients with cholangiocarcinoma is about 5-10%. Only 30%-40% of patients have the opportunity to obtain radical surgery. Surgical resection is limited by the extent of tumor spread along the bile duct branches and segments, and the degree of involvement of the portal vein and (or) hepatic artery branches. Complete resection with negative margins (R0) is the only possible radical treatment. Only 60%-78% of radical surgery for cholangiocarcinoma are considered to achieve true R0 resection, and the tumor-free margin is often very short. Even after R0 resection, the recurrence rate is as high as 50%-76%. Photodynamic therapy is a tumor specific ablation method with small side effects and repeated treatments will not produce drug resistance. It provides a new prospect for the treatment of cholangiocarcinoma. For the current patients with locally advanced cholangiocarcinoma, neoadjuvant photodynamic therapy is used to make them resectable. Demotion and subsequent resection may potentially improve their results. Similarly, patients with resectable margins can benefit from tumor downgrading by increasing their chances of undergoing R0 resection. In order to increase the negative rate of resection margins, and to ensure sufficient tumor-free margins of the bile duct stumps, the research is still blank. For patients with locally advanced cholangiocarcinoma with resectable margins, patients who meet the selection criteria are randomly divided into two groups A and B. Group A: neoadjuvant PDT therapy combined with radical surgery; Group B: radical surgery. This study aims to explore the clinical effectiveness and safety of neoadjuvant photodynamic therapy, as well as its role in destroying local tumors and enhancing systemic inflammation.This study plans to enroll 50 patients. It is planned to complete the enrollment operation within 2 years, and the follow-up observation will be continued for 5 years after the operation. All patients are expected to complete neoadjuvant PDT treatment and radical surgery within 2 years, survival period (5 years survival rate), R0 resection rate and local recurrence rate are the main observation indicators, and the bilirubin level, the number of intraoperative freezing, the length of the tumor-free margin of the tumor tissue, and the incidence of complications (biliary leakage, cholangitis, phototoxicity) are the secondary observation indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 to 75 years;
* Patients'gender was not limited;
* Patients with locally advanced cholangiocarcinoma who have a clear diagnosis of the primary disease and require surgical resection or potential surgical resection;
* No history of radiotherapy and chemotherapy;
* Willing to accept this clinical trial, sign informed consent and be able to cooperate with follow-up.

Exclusion Criteria:

* Women during pregnancy or breastfeeding, and those with mental illness;
* Patients allergic to porphyrin drugs, porphyria;
* Long-term use of glucocorticoids or autoimmune suppression;
* Surgical contraindication, including:

Child-Pugh C with hepatic encephalopathy Anyone with heart, lung, kidney dysfunction or other organ dysfunction, and cannot tolerate surgery.Hepatic ducts stone disease, who was diagnosed as Acute Cholangitis of Severe Type, especially complicated with bacteremia or septic shock. End stage disease, complicated with biliary cirrhosis or portal hypertension.Patients with long- term obstructive jaundice, dehydration, electrolyte disturbance or coagulation defects; Patients have the tendency or history of bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | During operation
  Compare the incidence of positive margins of bile duct after surgical resection of cholangiocarcinoma between the two groups
Local recurrence rate | 1-year post operation
  Compare the local recurrence rate of cholangiocarcinoma between the two groups
Survival time | 5-year post operation
  Compare the 5-year survival time of the two groups

SECONDARY OUTCOMES:
Bilirubin level | 1,3,6,12-month post operation
  Compare the Bilirubin level of the two groups
Complication rate | 1, 2,3,4,5,6,7,8-week Post operation
  Compare the incidence of bile leakage, cholangitis, phototoxicity and other complications between the two groups
Tumor-free margin length | During operation
  Compare the length of the tumor-free margin of the two groups of cholangiocarcinoma tissues

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lv, MD,PHD, Principal Investigator — China, Shaanxi First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- Yi Lv, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiedmann M, Caca K, Berr F, Schiefke I, Tannapfel A, Wittekind C, Mossner J, Hauss J, Witzigmann H. Neoadjuvant photodynamic therapy as a new approach to treating hilar cholangiocarcinoma: a phase II pilot study. Cancer. 2003 Jun 1;97(11):2783-90. doi: 10.1002/cncr.11401. PMID 12767091
- [Background] Wagner A, Wiedmann M, Tannapfel A, Mayr C, Kiesslich T, Wolkersdorfer GW, Berr F, Hauss J, Witzigmann H. Neoadjuvant Down-Sizing of Hilar Cholangiocarcinoma with Photodynamic Therapy--Long-Term Outcome of a Phase II Pilot Study. Int J Mol Sci. 2015 Nov 6;16(11):26619-28. doi: 10.3390/ijms161125978. PMID 26561801